CLINICAL TRIAL: NCT07309016
Title: The Effect of a Weighted Blanket on Lower Leg Cramps, Sleep Quality, Anxiety, and Stress in Pregnant Women: A Randomized Controlled Trial
Brief Title: Weighted Blanket in Pregnancy
Acronym: Weighted
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Serap Ejder Apay, Professor of Midwifery and Head of the Department of Midwifery, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/t
Record Dates: First submitted 2025-11-17; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Leg Cramps, Nocturnal; Poor Sleep Quality; Pregnancy; Anxiety; Stress
Keywords: Weighted blanket; sleep; anxiety; stress; cramps; pregnancy
MeSH Terms: conditions — Sleep-Wake Transition Disorders; Anxiety Disorders; Muscle Cramp

STUDY DESIGN:
Intervention Model Description: The study will be conducted using a single-group self-controlled design. Participants will first receive standard prenatal care without intervention for two weeks, followed by the weighted blanket intervention for two weeks. This approach allows comparison within the same individual, minimizing variability caused by personal differences or environmental factors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- This is a self-controlled randomized study. (Other): This study is designed to evaluate the effect of weighted blankets on lower leg cramps, sleep quality, anxiety and stress in pregnant women, assessing both the control group and the intervention group. This study is planned as a randomised self-controlled trial. This method was specifically chosen for the study design. The single-group approach allows for comparisons within each individual, significantly reducing the impact of personal differences. This minimises any bias that may arise from inter-individual variability. Furthermore, as multidimensional variables such as the lifestyle habits of pregnant women, their level of physical activity, dietary patterns, and environmental factors affecting sleep patterns have the potential to obscure the results of the study, this method aims to minimise the impact of these factors.
  Interventions: Device: Weighted Blanket

INTERVENTIONS:
Device: Weighted Blanket — The intervention involves the use of a weighted blanket designed to provide deep pressure stimulation during sleep. Each participant will first complete a 2-week control period with routine sleep conditions, during which baseline data will be collected. Immediately following this phase, participants will use the weighted blanket nightly for 2 weeks. No wash-out period will be applied between phases. Outcomes such as lower leg cramps, sleep quality, anxiety, and stress levels will be assessed and compared between the control and intervention periods within the same participants.

SUMMARY:
Pregnancy is frequently accompanied by sleep disturbances, musculoskeletal discomfort, anxiety, and stress, which may negatively affect maternal well-being and daily functioning. Weighted blankets, which provide deep pressure stimulation, have been used as a non-pharmacological method to promote relaxation, improve sleep quality, and reduce stress and anxiety. However, their effects have not been evaluated in pregnant women. This study aims to examine the effect of weighted blanket use on lower leg cramps, sleep quality, anxiety, and stress levels among pregnant women. The trial uses a randomized, self-controlled design in which each participant completes a 14-day control period without the blanket and a subsequent 14-day intervention period using the weighted blanket. Data will be collected using validated measurement tools. The findings are expected to provide evidence for a safe, non-pharmacological supportive approach that may enhance comfort and psychological well-being during pregnancy.

DETAILED DESCRIPTION:
Pregnancy involves physiological and psychological changes that may contribute to sleep difficulties, lower extremity cramping, and increased levels of anxiety and stress. Because pharmacological approaches are often limited during pregnancy, non-pharmacological strategies are important for promoting maternal comfort and well-being. Weighted blankets provide evenly distributed pressure across the body, generating deep pressure stimulation that may induce relaxation, reduce arousal, and support more stable sleep patterns.

This study is designed as a randomized, self-controlled trial to evaluate the effects of weighted blanket use on sleep quality, lower leg cramps, anxiety, and stress in pregnant women. The study includes one group of participants who undergo two consecutive phases:

Control Phase (14 days): Participants complete daily sleep diaries and standardized assessments without using a weighted blanket.

Intervention Phase (14 days): Participants receive an 8-kg glass-bead weighted blanket and use it during the sleep initiation period (approximately 40 minutes each night). Daily sleep diaries and standardized assessments are repeated following the intervention.

To support participant safety, the blanket weight will not exceed 8-10% of body weight, and participants will be instructed to use the blanket only during sleep onset. Participants will receive guidance on maintaining a safe sleep posture, particularly the left lateral position. Weekly follow-up phone calls will be conducted to monitor adherence, comfort, and potential adverse effects.

Hygiene measures include individual duvet covers for each participant, laundering of blankets between uses, and supervised storage of materials. All assessments will be administered by trained research personnel in accordance with standardized procedures.

Statistical analysis will include descriptive statistics, normality assessment, repeated-measures tests, and effect size calculations appropriate for within-subject comparisons. The study aims to determine whether weighted blanket use produces measurable improvements in sleep parameters, musculoskeletal discomfort, and psychological well-being during pregnancy. The results may contribute to evidence-based, complementary care practices in midwifery and prenatal health.

ELIGIBILITY:
Inclusion Criteria:

* Primarily pregnant women between the ages of 18 and 40 ,
* Low BMI (to be able to use 8kg weighted blanket),
* Gestational week ≥ 28,
* Third trimester pregnant women,
* Singleton pregnancy,
* Ability to communicate verbally and in writing in Turkish,
* Willingness to participate in research and comply with intervention protocols..

Exclusion Criteria:

* Those who have been diagnosed with high-risk pregnancy,
* Preeclampsia or eclampsia, placenta previa,
* Gestational diabetes requiring insulin,
* Diagnosis of fetal growth retardation,
* Polyhydramnios or oligohydramnios, asthma , sleep apnea or serious heart/circulatory problems,
* History of bleeding during pregnancy,
* Obstetric complications requiring close medical monitoring.
* Multiple pregnancies,
* Previously diagnosed with a sleep disorder,
* Having been diagnosed with a psychiatric disorder
* Multiparous pregnant women,
* Pregnant women in the first two trimesters ,
* Night shift workers

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index - PSQI | Baseline (Day 0-14; control phase) Post-intervention (Day 15-28; after weighted blanket use)
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index, a validated 19-item instrument that generates a total score based on seven components of sleep. Total PSQI scores range from 0 to 21, with higher scores indicating poorer sleep quality. The change in PSQI total score from baseline (control period) to post-intervention will be evaluated.
Leg Cramp Questionnaire Form | Baseline (Day 0-14; control phase) Post-intervention (Day 15-28)
  Lower leg cramps will be evaluated using participant-reported frequency (number of cramps per week) and severity (rated on a 0-10 Numeric Rating Scale, where 0 = no pain and 10 = most severe pain). Changes between the 14-day control phase and the 14-day intervention phase will be assessed.
Perinatal Anxiety Screening Scale (PASS) | Baseline (after 14-day control phase) Post-intervention (after 14 days of weighted blanket use)
  Anxiety levels will be assessed using the Perinatal Anxiety Screening Scale, a validated 31-item instrument. The total PASS score ranges from 0 to 93, with higher scores indicating greater perinatal anxiety. Total scores will be compared before and after the intervention.
Pregnancy Stress Rating Scale | Baseline (after 14-day control phase) Post-intervention (after 14 days of weighted blanket use)
  Pregnancy-related stress will be measured using the Pregnancy Stress Rating Scale, a validated 36-item scale. Total scores range from 0 to 144, with higher scores reflecting higher levels of pregnancy-related stress. The change in PSRS total score from baseline to post-intervention will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Serap EJDER APAY, Professor, Principal Investigator — Atatürk University Faculty of Health Sciences, Department of Midwifery
Locations (1):
- Atatürk University Instiute of Health Sciences, Department of Midwifery, Erzurum, Lütfen Seçiniz., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves a limited number of participants and data contain potentially identifiable information. Only summarized results will be made available upon reasonable request.